CLINICAL TRIAL: NCT03925662
Title: Clinical Study Evaluating Mebendazole as Adjuvant Therapy in Patients With Colorectal Cancer
Brief Title: Mebendazole as Adjuvant Treatment for Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: colon cancer
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Bevacizumab; Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folfox with avastin (Active Comparator): Folfox with avastin only
  Interventions: Drug: Folfox with avastin
- Mebendazole (Experimental): Folfox with avastin with mebendazole
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Folfox with avastin — Folfox with avastin only
  Other Names: folfox 4
  Arms: Folfox with avastin
Drug: Mebendazole — Folfox with avastin with mebendazole
  Other Names: mebendazol
  Arms: Mebendazole

SUMMARY:
mebendazole treating colon cancer

DETAILED DESCRIPTION:
mebendazole as adjuvant treatment for colon cancer

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer stage 4.

Exclusion Criteria:

* Agranulocytosis
* Pregnancy
* Allergy to mebendazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with tumour response | 6 months
  number of patients with response

CONTACTS AND LOCATIONS:
Overall Officials: Reham El-ghoneimy, Msc, Principal Investigator — Tanta University - Faculty of Pharmacy; Sahar Hegazy, Prof, Principal Investigator — Tanta University - Faculty of Pharmacy; Gamal el-azab, Prof, Study Director — Tanta University - Faculty of Pharmacy; Fatma Zakaria, Prof, Study Chair — Tanta University
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hegazy SK, El-Azab GA, Zakaria F, Mostafa MF, El-Ghoneimy RA. Mebendazole; from an anti-parasitic drug to a promising candidate for drug repurposing in colorectal cancer. Life Sci. 2022 Jun 15;299:120536. doi: 10.1016/j.lfs.2022.120536. Epub 2022 Apr 3. PMID 35385794